CLINICAL TRIAL: NCT04727606
Title: Research Project: Pilot Study on Oral Urea Use in Patients at High Risk of Kidney Stone Recurrence
Acronym: Ure-Na
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: We never got Health Canada approval
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20.259
Record Dates: First submitted 2020-11-17; First posted 2021-01-27 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open label (Experimental): The study provides for a single group, which will be its own control (pre/post intervention study). Participants in the study will receive Oral Urea (Ure-Na) treatment at a dose of 30 grams per day (2 x 15 gram pouches per day) for 1 month
  Interventions: Drug: Ure-Na

INTERVENTIONS:
Drug: Ure-Na — * Participants in the study will receive Oral Urea (Ure-Na) treatment at a dose of 30 grams per day (2 x 15 gram pouches per day)
  * Treatment will continue for approximately 1 month.

SUMMARY:
In clinical practice, many patients are not able to modify their habits to achieve a high level of diuresis and fluid intake and therefore are at an elevated risk for stone recurrence.

The investigators think that Ure-Na (osmotic agent) taking could help to increase urine volume and decrease urine concentration, which would be of benefit in the prevention of kidney stones.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years of age
* High risk for recurrence (1 or more of) Bilateral or complex stones, Recurrent stones, Family history (1st degree relative), Non-calcium stones, Solitary kidney or anatomical abnormality, Nephrocalcinosis, Systemic disease with risk of stones (tubular acidosis, cystinuria, etc.)
* Diuresis < 1.8 L/24 hours despite recommendations from physicians and/or nutritionist at the kidney stone clinic (as documented in the previous 6 months)

Exclusion Criteria:

* Patient does not meet 1 of the 3 inclusion criteria
* Pregnancy or breastfeeding
* Lack of understanding about the protocol and effects of Ure-Na
* Expected inability to adequately increase fluid intake on Ure-Na

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in urine output at 1 week and 1 Month | 1 week and 1 month
  variation in 24-hour diuresis and urine biochemistry

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dion M, Ankawi G, Chew B, Paterson R, Sultan N, Hoddinott P, Razvi H. CUA guideline on the evaluation and medical management of the kidney stone patient - 2016 update. Can Urol Assoc J. 2016 Nov-Dec;10(11-12):E347-E358. doi: 10.5489/cuaj.4218. Epub 2016 Nov 10. No abstract available. PMID 28096919
- [Background] Borghi L, Meschi T, Amato F, Briganti A, Novarini A, Giannini A. Urinary volume, water and recurrences in idiopathic calcium nephrolithiasis: a 5-year randomized prospective study. J Urol. 1996 Mar;155(3):839-43. PMID 8583588
- [Background] Soupart A, Coffernils M, Couturier B, Gankam-Kengne F, Decaux G. Efficacy and tolerance of urea compared with vaptans for long-term treatment of patients with SIADH. Clin J Am Soc Nephrol. 2012 May;7(5):742-7. doi: 10.2215/CJN.06990711. Epub 2012 Mar 8. PMID 22403276
- [Background] Berl T. Impact of solute intake on urine flow and water excretion. J Am Soc Nephrol. 2008 Jun;19(6):1076-8. doi: 10.1681/ASN.2007091042. Epub 2008 Mar 12. PMID 18337482
- [Background] Decaux G, Brimioulle S, Genette F, Mockel J. Treatment of the syndrome of inappropriate secretion of antidiuretic hormone by urea. Am J Med. 1980 Jul;69(1):99-106. doi: 10.1016/0002-9343(80)90506-9. PMID 7386514
- [Background] Verbalis JG, Baldwin EF, Neish PN, Robinson AG. Effect of protein intake and urea on sodium excretion during inappropriate antidiuresis in rats. Metabolism. 1988 Jan;37(1):46-54. doi: 10.1016/0026-0495(88)90028-5. PMID 3336285
- [Background] Nayan M, Elkoushy MA, Andonian S. Variations between two 24-hour urine collections in patients presenting to a tertiary stone clinic. Can Urol Assoc J. 2012 Feb;6(1):30-3. doi: 10.5489/cuaj.11131. PMID 22396364